## Effects of High-Intensity Interval Training and Strength Training On Levels of Testosterone and Physical Activity among Women with Polycystic Ovary Syndrome.

ClinicalTrials registration no: NCT04942366

**Date: 9-March-2021** 

## **Statistical Analytical Plan:**

For the analysis, the data was entered and analyzed in MedCalc software version 19.0.5. Descriptive statistics were performed for demographic information and this data is presented in terms of frequency and percentage. Shapiro-Wilk test was used to determine the normality of data.

**For BMI:** Shapiro-Wilk test was used to determine the normality of data and the data was normally distributed so paired T-test was performed for within group analysis. Independent T-test was performed for the comparison between the two groups.

**For Serum testosterone:** Shapiro-Wilk test was used to determine the normality of data and the data was normally distributed so paired T-test was performed for within group analysis. Independent T-test was performed for the comparison between the two groups.

**For Body fat percentage:** Shapiro-Wilk test was used to determine the normality of data. The data was not normally distributed so, Wilcoxon sign rank test was performed for within group analysis. Independent T-test was performed for the comparison between the two groups.

**For IPAQ:** Shapiro-Wilk test was used to determine the normality of data. The data was not normally distributed so, Wilcoxon sign rank test was performed for within group analysis. Independent T-test was performed for the comparison between the two groups.